CLINICAL TRIAL: NCT01474720
Title: Immunologic Response to Varicella Zoster Vaccination With Zostavax in Patients With Systemic Lupus Erythematosus
Brief Title: Zostavax in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oklahoma Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OMRF 11-45
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2011-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Lupus; SLE; Zostavax; shingles
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SLE patients (Experimental): Subjects with mild SLE over age 50 years will receive open-label Zostavax vaccine.
  Interventions: Drug: Zostavax vaccine
- Healthy subjects (Active Comparator): Healthy subjects aged 50 years and older without any history of autoimmune disease will receive zostavax vaccine. Immune responses to varicella zoster virus and adverse events will be compared to those seen in SLE patients
  Interventions: Drug: Zostavax vaccine

INTERVENTIONS:
Drug: Zostavax vaccine — Commercially available Zostavax vaccine will be administered subcutaneously according to package insert guidelines. Each 0.65-mL dose contains a minimum of 19,400 PFU (plaque-forming units) of Oka/Merck strain of VZV.

SUMMARY:
Individuals with systemic lupus erythematosus (SLE, lupus) appear to be at increased risk for the development of shingles, a painful reactivation of the varicella zoster virus that causes chicken pox.

The investigators propose to study the immune response to commercially available Zostavax vaccine (shingles vaccine) in adult patients with SLE who have minimal disease activity and are on mild immunosuppressant medications, and to compare the immune response to that seen in healthy people following vaccination. Acceptable immunosuppressive drugs permitted in the study are those felt to be safe according to Centers for Disease Control guidelines.

Ten healthy people and 10 SLE patients (all over 50 years of age) will be recruited to receive a single, standard dose of Zostavax. Blood samples and physical examination will be performed prior to injection, then 2,6,and 12 weeks following vaccination. All participants will receive active vaccine, there is no placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Willing and able to provide written informed consent
* History of primary varicella vaccination or positive VZV IgG antibodies
* Diagnosis of SLE according to ACR criteria for > 1 year; or healthy control subject
* Stable, mild disease activity as defined by a clinical SLEDAI score ≤ 4
* Current medical treatment for SLE has been stable for 4 weeks prior to screening
* Acceptable immunosuppressive medications are limited to
* Prednisone ≤ 10 mg daily
* Methotrexate ≤ 20 mg weekly
* Azathioprine ≤ 150 mg daily
* Hydroxychloroquine ≤ 6.5 mg/kg daily
* Female subjects of childbearing potential and non-sterile males must agree to use acceptable form of contraception for the duration of the study

Exclusion Criteria:

* History of receiving any VZV-containing vaccine (primary varicella or zoster)
* History of herpes zoster reactivation within 5 years prior to enrollment
* Received any live vaccine within 6 weeks or inactivated/recombinant vaccine within 2 weeks of enrollment
* Known Hepatitis B, C or HIV virus infection
* History of drug or alcohol abuse within 1 year of screening
* Rituximab therapy within 2 years of screening
* Cyclophosphamide within 6 months of screening
* Biologic therapy (TNF inhibitors, CTLA-4Ig, etc.) within 6 months of screening
* Use of mycophenolate mofetil within 3 months of screening
* History of receiving immunoglobulin or other blood product within 3 months of screening
* Allergic reaction, intolerance or other contraindication to use of famciclovir.
* Has received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 3 months of screening; or expects to receive another experimental/investigational agent within 6 months post immunization.
* Pregnant or lactating women
* Unwilling to use acceptable method of contraception for the duration of the study
* WBC <3.0; ANC <1500; CD4+ <200
* Proteinuria >1.5 mg/day
* Impaired renal function defined by serum Cr >1.5
* Transaminases > 2x upper limit of normal
* Clinical SLEDAI > 4
* Active lupus nephritis or cerebritis
* History of neoplastic disease within 5 years of screening, except for completely excised non-melanoma cancer of the skin or in-situ carcinoma of the uterine cervix.
* History of any hematological malignancy, current bleeding disorder or taking anticoagulant medication (heparin or warfarin).
* Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Has a moderate to severe acute illness and/or oral temperature greater or equal to 100.0oF, within 72 hours prior to vaccination (this may result in temporary delay of vaccination).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Cell-mediated immune response to varicella at 12 weeks following vaccination | 12 weeks
  Peripheral blood will be drawn at baseline, then at 2,6, and 12 weeks following vaccination. Peripheral blood mononuclear cells will be assessed for measures of varicella-zoster specific immunity.

SECONDARY OUTCOMES:
Antibody response to Zostavax vaccination | 12 weeks
  Varicella specific IgG antibodies will be compared between baseline and 12 weeks post vaccination.
Adverse events | 12 weeks
  The development of adverse events, particularly injection site reactions or rash near the injection site will be tabulated and compared between SLE and healthy control groups

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Guthridge JM, Cogman A, Merrill JT, Macwana S, Bean KM, Powe T, Roberts V, James JA, Chakravarty EF. Herpes zoster vaccination in SLE: a pilot study of immunogenicity. J Rheumatol. 2013 Nov;40(11):1875-80. doi: 10.3899/jrheum.130170. Epub 2013 Sep 15. PMID 24037550